CLINICAL TRIAL: NCT07169214
Title: Evaluation of Safety, Efficacy, and Pharmacokinetics of BT-114143 Injection in Patients With Abnormal Uterine Bleeding
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ScinnoHub Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT-114143-I-02
Record Dates: First submitted 2025-08-14; First posted 2025-09-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Abnormal Uterine Bleeding
MeSH Terms: conditions — Metrorrhagia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- low-dose group (Experimental): Subjects received low-dose BT-114143 Injection treatment
  Interventions: Drug: BT-114143 Injection at low dose
- Medium-dose group (Experimental): Subjects received Medium-dose BT-114143 Injection treatment
  Interventions: Drug: BT-114143 Injection at Medium-dose
- High-dose Group (Experimental): Subjects received High-dose BT-114143 Injection treatment
  Interventions: Drug: BT-114143 Injection at High-dose
- control group (Placebo Comparator): The subjects receive normal saline treatment.
  Interventions: Drug: control group

INTERVENTIONS:
Drug: BT-114143 Injection at low dose — A total of 10 subjects were enrolled. All of them received BT-114143 Injection at low dose. BT-114143 will be administered twice daily for three consecutive days.
  Arms: low-dose group
Drug: BT-114143 Injection at Medium-dose — A total of 10 subjects were enrolled. All of them received BT-114143 Injection at Medium-dose. BT-114143 will be administered twice daily for three consecutive days.
  Arms: Medium-dose group
Drug: BT-114143 Injection at High-dose — A total of 10 subjects were enrolled. All of them received BT-114143 Injection at High-dose. BT-114143 will be administered twice daily for three consecutive days.
  Arms: High-dose Group
Drug: control group — The ratio of subjects in the experimental group to those in the control group is 10:3, with 3 placebo - treated control subjects corresponding to each dose group. The subjects will receive placebo treatment twice a day for 3 consecutive days.
  Arms: control group

SUMMARY:
This is a randomized, double-blind, placebo-controlled, multiple-dose escalation, Phase Ib clinical study conducted in patients with abnormal uterine bleeding (e.g., AUB). It aims to evaluate the safety, efficacy, pharmacokinetic characteristics of multiple administrations of BT-114143 Injection at different doses, as well as to explore changes in coagulation-related biomarkers and quality of life.

It is planned to enroll 39 adult patients with abnormal uterine bleeding.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to sign the informed consent form before any study-related procedures are performed, and be willing and able to comply with the study requirements;
2. Premenopausal female subjects, aged 18-50 years, including 18 and 50 years;
3. Have regular menstrual cycles in the past 6 months, with a menstrual cycle of ≥21 days and ≤35 days, and a menstrual period duration of ≤14 days;
4. Meet the diagnosis of abnormal uterine bleeding and agree to be admitted for treatment. Assessed by the alkaline hemoglobin method, in 2 consecutive menstrual cycles during the screening period, the menstrual blood loss is >80 ml in both cycles; or the blood loss in any one cycle is ≥160 ml;
5. The pregnancy test result is negative before randomization;
6. Those with a body mass index [BMI = weight (kg) / height² (m²)] of 18.5-28.0 kg/m² (including the boundary values).

Exclusion Criteria:

1. Patients with known endometrial polyps > 1.5 cm, endometrial malignancy, or atypical hyperplasia;
2. Patients with known or investigator-determined ovulatory dysfunctional abnormal uterine bleeding who require hormonal therapy;
3. Patients identified by investigators as having iatrogenic abnormal uterine bleeding;
4. Patients with abnormal uterine bleeding related to coagulation dysfunction, including but not limited to those with laboratory test results showing: platelet count ≤ 100×10⁹/L, or APTT prolonged by ≥ 10s beyond the upper limit of normal, or PT prolonged by ≥ 3s beyond the upper limit of normal;
5. Patients with bleeding caused by cervical or vaginal lesions;
6. Patients who have undergone major surgery within 6 months prior to screening;
7. Patients determined by investigators before randomization to require surgical treatments such as total hysterectomy, myomectomy, hysteroscopic treatment, uterine artery embolization, or ablation during the study period;
8. Patients who have received the following medications within 3 months prior to randomization: gonadotropin-releasing hormone agonists; sex hormone drugs administered orally, by injection, vaginally, or transdermally (including but not limited to drugs containing estrogen or progesterone); selective estrogen receptor modulators; hormonal intrauterine devices (LNG-IUS). For long-acting (3-month) gonadotropin-releasing hormone agonists or progesterone preparations, the last administration must be no later than 6 months prior to randomization;
9. Patients who have used danazol, desmopressin, tranexamic acid, aminocaproic acid, or traditional Chinese medicines for the treatment of menorrhagia within 3 months prior to randomization;
10. Patients who need to receive anticoagulants (e.g., warfarin, heparin, etc.) or antiplatelet therapies (e.g., clopidogrel, ticagrelor, etc.) during the study period;
11. Patients with intolerance or contraindications to BT-114143 Injection;
12. Patients who have participated in clinical trials of other investigational drugs, biological agents, or medical devices and received therapeutic interventions within 30 days prior to screening;
13. Patients with clinically severe diseases such as known disorders of the circulatory, endocrine, nervous, digestive, respiratory, urinary, hematological, immunological, psychiatric, or metabolic systems, as assessed by investigators as unsuitable for participation in the trial;
14. Patients with a known history of glaucoma or retinopathy, as assessed by investigators as unsuitable for participation in the trial;
15. Untreated or poorly controlled thyroid dysfunction, except for mild subclinical hypothyroidism (i.e., TSH < 10 mIU/L with normal FT4 and TT4);
16. Patients with a known history of thrombotic diseases, including but not limited to pulmonary embolism, deep vein thrombosis, etc.;
17. Patients diagnosed with malignant tumors within the past 5 years, except for cured basal cell carcinoma of the skin;
18. Patients with cervical cytology results indicating a risk of cervical cancer within 1 year prior to the screening period and requiring treatment.
19. Patients with one or more of the following abnormal laboratory test results before randomization:

    * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 1.5 × ULN;
    * Total bilirubin > 1.5 × ULN, except for patients with Gilbert's syndrome;
    * eGFR ≤ 60 mL/min/1.73 m² (calculated using the CKD-EPI formula);
    * Hemoglobin < 90 g/L;
20. Patients with known infection of human immunodeficiency virus (HIV), or positive hepatitis B surface antigen (HBsAg), or positive hepatitis C virus antibody (HCV Ab);
21. Alcohol abusers (i.e., consuming more than 14 standard units of alcohol per week within 3 months before screening (1 standard unit contains 14g of alcohol, such as 360ml of beer, 45ml of spirits with 40% alcohol content, or 150ml of wine)), or those with a history of drug abuse (such as morphine, tetrahydrocannabinolic acid, methamphetamine, 3,4-methylenedioxymethamphetamine, ketamine) within 1 year before screening, or with mental or neurological diseases that investigators consider may affect participation in the study;
22. Pregnant or lactating women, or subjects who had unprotected sex within 14 days before screening;
23. Subjects who have plans for pregnancy from the time of signing the informed consent form until 3 months after the last administration, or subjects (or their partners) who are unwilling to take effective contraceptive measures (specific contraceptive measures are shown in Appendix 1);
24. Patients with any condition or result that investigators or designated personnel consider may pose a risk to subjects or the implementation of the study;

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-09-23 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
safety evaluation | from the first administration to 2 weeks after the last administration
  The incidence of abnormal laboratory values, clinically significant physical examination findings, vital signs, electrocardiograms (ECGs), and/or treatment-related adverse events/serious adverse events.

SECONDARY OUTCOMES:
Change of menstrual bleeding volume from baseline | from signing the informed consent to 2 weeks after the last administration
  Sanitary products used by subjects are collected regularly, and menstrual blood loss is measured by the alkaline hemoglobin method.
Percentage change of menstrual bleeding volume from baseline | from signing the informed consent to 2 weeks after the last administration
  Sanitary products used by subjects are collected regularly, and menstrual blood loss is measured by the alkaline hemoglobin method.
The difference in the number of menstrual bleeding days between the post-treatment period and the baseline period in subjects. | From signing the informed consent to 2 weeks after the last administration
The proportion of subjects with menstrual blood loss ≤ 80 ml after treatment. | from signing the informed consent to 2 weeks after the last administration
The proportion of subjects with a reduction in menstrual blood loss of ≥50 ml after treatment compared with the baseline | from signing the informed consent to 2 weeks after the last administration
The proportion of subjects with a reduction in menstrual blood loss of ≥36 ml after treatment compared with the baseline. | from signing the informed consent to 2 weeks after the last administration
The change in the Menorrhagia Impact Questionnaire (MIQ) score from baseline after treatment in subjects. | from signing the informed consent to 2 weeks after the last administration
  Evaluate Menorrhagia Impact Questionnaire (MIQ) score at screening visit and treatment period. The MIQ consists of six individual measures or items. The first 4 items are evaluated by using 4-point (item 1) or 5-point (items 2-4) response scales. No summative scale is derived for item 5 as it serves as a descriptive tool to characterize limitations of specific activities. Item 6 represents a global assessment (impact, degree, and meaningfulness) of the change in MBL when compared to the previous period. Scores correlate with symptom severity; a higher score indicates more severe heavy menstrual bleeding.
The change in the Menstrual Discomfort Questionnaire (MDQ) score from baseline after treatment in subjects. | from signing the informed consent to 2 weeks after the last administration
  A total of 46 related items that reflect eight subscales were included in the MDQ. Each of the eight subscales is composed of an interrelated set of items, and each item is scored on a 5-point Likert scale. The scale ranges from 0 to 184, with higher scores indicating more severe heavy menstrual bleeding.

OTHER OUTCOMES:
To characterize the pharmacokinetic (PK) profile of BT-114143 | Three days after administration
  Plasma concentration of BT-114143 will be measured and following PK parameters will be characterized: Maximum observed concentration (Cmax); Time to Cmax (Tmax); area under the plasma concentration-time curve (AUC) from the time 0 to the last quantifiable time point (AUC0-t); AUC from the time 0 to infinity (AUC0-inf); half-life (t1/2); apparent clearance (CL/F); apparent volume of distribution (Vz/F)
Changes in Plasminogen Activity Results from Baseline | Three days after administration
  Blood samples will be collected to determine the changes in plasminogen activation over time.
Prothrombin Time（PT） | Three days after administration
  The change of PT from baseline
Activated Partial Thromboplastin Time（APTT） | 3 days after administration
  The change in Activated Partial Thromboplastin Time (APTT) from baseline
International Normalized Ratio（INR） | 3 days after administration
  The change in INR (International Normalized Ratio) from baseline
Thrombin Time（TT） | 3 days after administration
  The change in TT (Thrombin Time) from baseline
Fibrinogen（FIB） | 3 days after administration
  The change in FIB (Fibrinogen) from baseline
D-Dimer | 3 days after administration
  The change in D-Dimer (D-Dimer) from baseline
Changes in Thromboelastography (TEG) Parameters | 3 days after administration
  Blood samples will be collect at each timepoints and TEG parameter (including R, K, Angle, MA, LY30, and CI values) will be measured to determine coagulation function of each subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No